CLINICAL TRIAL: NCT05408884
Title: Miracle Friends and Miracle Money Evaluation
Brief Title: Miracle Messages Evaluation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Southern California (Other)
Collaborators: Miracle Messages (Unknown)
Responsible Party: Principal Investigator, Benjamin F. Henwood, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UP-22-00242
Record Dates: First submitted 2022-05-26; First posted 2022-06-07 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Homelessness

STUDY DESIGN:
Who Masked: Participant
Masking Description: Those assigned to the Miracle Money condition are not notified that they have been selected to receive monthly income until after they have actively engaged in the Miracle Friends intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Miracle Friends (Active Comparator): Participants selected to receive a social support "phone buddy" program.
  Interventions: Other: Social Support
- waitlist (No Intervention): Waitlisted for the social support "phone buddy" program.
- Miracle Money (Experimental): Participants who receive $750 monthly income for 12 months based on having engaged in the Miracle Friends program
  Interventions: Other: Social Support; Other: Basic income

INTERVENTIONS:
Other: Social Support — Social support "phone buddy" program.
  Other Names: Miracle Friends
  Arms: Miracle Friends; Miracle Money
Other: Basic income — $750 per month for 12 months
  Other Names: Miracle Money
  Arms: Miracle Money

SUMMARY:
The project will conduct a randomized control trial (RCT) of an innovative program for people experiencing homelessness (PEH) that initially designed to address social isolation and loneliness among people experiencing homelessness but subsequently paired with an economic poverty-reduction intervention. The social support intervention, known as "Miracle Friends," pairs an unhoused person with a volunteer "phone buddy." The poverty reduction intervention, known as "Miracle Money," provides guaranteed basic income of $750 per month for 1 year to Miracle Friends participants.

DETAILED DESCRIPTION:
The project will conduct a randomized control trial (RCT) of an innovative program for people experiencing homelessness (PEH) that initially designed to address social isolation and loneliness among people experiencing homelessness but subsequently paired with an economic poverty-reduction intervention. The social support intervention, known as "Miracle Friends (MF)," pairs an unhoused person with a volunteer "phone buddy." The poverty reduction intervention, known as "Miracle Money (M$)," provides guaranteed basic income of $750 per month for 1 year to MF participants. The RCT will have 3 arms of PEH who expressed interest in the phone buddy program: (1) those assigned to Miracle Friends; (2) those assigned to Miracle Money, which is not disclosed until after they actively engage in the Miracle Friends program; (3) And those assigned to a waitlist for Miracle Friends. To recruit for the study, the Miracle Friends program engage PEH through a variety of homeless services partners and introduce the MF program. Anyone who is interested in the MF program is provided information about a 15-month longitudinal study and referred to the research team to complete an eligibility screener. The research team explains the interview protocols that include receiving a $30 incentive each time a survey is completed that includes a baseline and 5 quarterly surveys. Participants will also be notified about being randomly selected to either be offered MF or put on a waitlist. Those assigned to the M$ are not notified about receiving monthly income until after they engage in the MF program. Information about frequency of contact with the MF social support volunteer and volunteer demographics will be provided directly from the Miracle Friends administrative data records.

ELIGIBILITY:
Inclusion Criteria:

* being 18 years old or older;
* speaks English;
* currently experiencing homelessness;
* has expressed interest in signing up for the Miracle Friends ("phone buddy") program.

Exclusion Criteria:

* not meeting the inclusion criteria;
* not able to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 759 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Homelessness/Housing status using questions from the Los Angeles Homeless Count | Measured quarterly for 15 months.
  In the past 30 days, please indicate all places where you have slept for at least one night: 1. My own apartment or home 2. Someone else's apartment or home 3. In a shelter, emergency, temporary housing, 4. Hotel/motel provided by an agency 5. Outside on the street, park, or beach 6. Tent or makeshift shelter 7. In a bus station, train station, airport 8. Abandoned building 9. In a vehicle (car, van, recreation vehicle (RV), truck) 10. An institution, hospital, or facility

SECONDARY OUTCOMES:
Employment status using questions from the Los Angeles Homeless Count | Measured quarterly for 15 months.
  What is your employment status?
  1. Employed, full-time (35 hours a week or more)
  2. Employed, part-time
  3. Unemployed, looking for work
  4. Unemployed, not looking for work
  5. Retired, receiving retirement benefits
  6. Retired, not receiving benefits
Health status using Patient-Reported Outcomes Measurement InformationSystem (PROMIS) Scale 1.2 | Measured quarterly for 15 months.
  In general, how would you rate your physical/mental health?
  1. Excellent
  2. Very good
  3. Good
  4. Fair
  5. Poor
University of California Los Angeles (UCLA) Loneliness Short Version | Measured quarterly for 15 months.
  3 item questionnaire: How often do you feel that you lack companionship?
  How often do you feel left out? How often do you feel isolated from others?
  1. Hardly ever
  2. Some of the time
  3. Often

CONTACTS AND LOCATIONS:
Overall Officials: Ben Henwood, PhD, Principal Investigator — University of Southern California
Locations (1):
- Miracle Messages, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Henwood BF, Kim BE, Stein A, Corletto G, Suthar H, Adler KF, Mazzocchi M, Ip J, Padgett DK. Miracle friends and miracle money in California: a mixed-methods experiment of social support and guaranteed income for people experiencing homelessness. Trials. 2024 Apr 29;25(1):290. doi: 10.1186/s13063-024-08109-6. PMID 38685123